CLINICAL TRIAL: NCT00915369
Title: A Multicentre Phase I Study Of Cremophor FreePaclitaxel Nanoparticle In Advanced Breast Cancer
Brief Title: A Clinical Trial to Study the Effects of Nanoparticle Based Paclitaxel Drug, Which Does Not Contain the Solvent Cremophor, in Advanced Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fresenius Kabi Oncology Ltd. (Industry)
Responsible Party: Dr. S. K. Mishra, Vice President - Clinical Research & Medical Services, Fresenius Kabi Oncology Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO/NDR/02/2008/01
Record Dates: First submitted 2009-06-03; First posted 2009-06-08 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nanoxel (Paclitaxel Nanoparticle formulation ) — Nanoxel (Nanoparticle Paclitaxel) at 4 different dose levels of 220, 260, 310 and 375 mg/m2. Each patient will recieve upto 6 cycles.

SUMMARY:
This study is a multicentre, open label, non-randomized phase I study. The main objectives of the study are to determine the pharmacokinetic profile of the drug at different dose levels in the patients with Advanced Breast Cancer. Maximum Tolerated Dose (MTD) and safety of Paclitaxel Nanoparticle will also be simultaneously assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histopathologically /cytologically confirmed advanced breast cancer, refractory / recurrent* to previous anthracycline treatment as adjuvant or first line therapy for metastasis.
* Patients with ER/PR -ve or ER/PR receptor status unknown (defined as no histopathological evidence for confirmation of ER/PR status)
* Patients must be of 18-65 years of age (inclusive of both)
* Patients with ECOG performance status between 0 - 2
* Patients with at least one measurable lesion as per RECIST

Exclusion Criteria:

* Patients with ER/PR positive status. Patients who demonstrate HER2 over expression will be excluded. Alternatively, the patients enrolled should have previously received trastuzumab. HER2 over expression should be demonstrated by IHC 3+, IHC 2+ or with FISH/CIS.
* Patients with known history of hypersensitivity to paclitaxel or any other taxane or compounds chemically / biologically related to paclitaxel or excipients.
* Patients requiring any concurrent chemotherapy, hormonal therapy immunotherapy, therapy with biologicals or radiotherapy for the disease. (Patients requiring local radiotherapy for non- target bone lesion will be included).
* Patients with known CNS lesions (brain metastasis or carcinomatous meningitis).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcomes of the study would be the Pharmacokinetic data at all the four dose levels (220, 260, 310 and 375 mg/m2); Ability to identify a dose higher than 220 mg/m2 that demonstrate better efficacy and manageable toxicity | Throughout the study

SECONDARY OUTCOMES:
evaluation of the effect of Paclitaxel Nanoparticle formulation on QTc. | Throughout the study

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Nizam'S Institute of Medical Sciences, Hyderabaad, Andhra Pradesh
  - Kidwai Memorial Institute of Oncology, Bangalore, Karnataka
  - SEAROC Cancer Center, S K Soni Hospital, Jaipur, Rajasthan